CLINICAL TRIAL: NCT03557723
Title: Effect of Art Museum Activity Program for the Elderly on Health: A Pilot Observational Study
Status: Completed | Type: Observational
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, Principal Investigator, Jewish General Hospital
Other Study IDs: CODIM-FLP-17-083
Record Dates: First submitted 2018-01-31; First posted 2018-06-15 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Health; Quality of Life; Social Interaction
Keywords: Community-dwellers,older adults, museum, art

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Art activities program — The intervention will be the MMFA art activities program "Les Beaux Jeudis". Three activities will be examined:
  1. Cultural mediation workshop
  2. Supervised visit and tour of the museum
  3. Cultural mediation workshop combined with supervised visit and tour of the museum
  The duration of the MMFA art activities program "Les Beaux Jeudis" will be 3 months. Each participatory-based art activity is a weekly activity.

SUMMARY:
Older adults, defined as 65 years or older, are increasing in number and representing a larger part of Canadian population. Assessing and addressing the needs of this growing number of individuals is essential. Practicing art and/or being involved in cultural programs could enhance health and quality of life of older adults. The overall objective of the proposal is to describe the characteristics (i.e.; socio-demographic, health condition and quality of life) and their changes in older adults participating in the Montreal Museum of Fine Arts (MMFA; Quebec, Canada) art activities program called "Les Beaux Jeudis". An observational, prospective, cohort study, before and after participation in MMFA art activities program "Les Beaux Jeudis" will be performed.

DETAILED DESCRIPTION:
The population is aging. Aging is often associated with worsening health, which increases the risk of a poor quality of life. It has been reported that practicing art and/or being involved in cultural programs, especially participatory-based art activities, enhances the quality of life of patients. No effect on health and quality of life has been reported in community-dwellers living independently at home. Since October 2015, the Montreal Museum of Fine Arts (MMFA; Quebec, Canada) has successfully initiated a series of participatory-based art activities called "Les Beaux Jeudis" for older community-dwellers. This art museum program includes several activities such as: cultural mediation workshops, supervised museum visit and tours as well as a combination of both activities. Here, the investigator has the unique opportunity to examine whether and how the MMFA art activities program influences health conditions and the quality of life in older community-dwellers.

Objectives

The objectives of the proposal are to examine: 1) The socio-demographic, health and quality of life characteristics of older adults before, during and after their participation in the MMFA art activities program "Les Beaux Jeudis" 2) Compliance to the MMFA art activities program 3) Self-assessment of health and quality of life feasibility using a personalized e-Health application, accessible online on the web platform of the Telehealth McGill integrated university health network.

Methods

The design of this study is: observational, prospective, cohort study, before and after participation in the MMFA art activities program "Les Beaux Jeudis". The recruited population will be older adults who are participants of the MMFA art activities program. Three participatory-based art activities are examined: 1) Cultural mediation workshop 2) Supervised museum visit and tour of museum 3) Cultural mediation workshop combined with supervised museum visit and tour of museum. Each participatory-based art activity is a weekly activity. The duration of the MMFA art activities program is 3 months. Five outcomes are examined: Socio-demographic characteristics, health condition, quality of life, compliance to the MMFA art activities program and the usability of a personalized e-Health application.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years and over
* Internet access with an electronic device (i.e.; laptop, computer, smartphone, tablet) at the participant's place of living

Exclusion Criteria:

* Individuals participating in cultural mediation workshop
* Individuals participating in supervised visit and tour of the museum
* Individuals participating in cultural mediation workshop combined with supervised visit and tour of the museum

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The recruited population will be older adults who are the participants of the Montreal Museum of Fine Arts activities program "Les Beaux Jeudis".
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2018-09-13 (Actual); Study Completion 2018-09-13 (Actual)

PRIMARY OUTCOMES:
Health | 3 months follow-up
  Using an electronic self-administered questionnaire

SECONDARY OUTCOMES:
Quality of life | 3 months follow-up
  Using the Warwick-Edinburg Mental Well-being scale.
  -Warwick-Edinburg Mental Well-being scale is a validated questionnaire composed by 14 positively worded item scale with five response categories. It covers most aspects of positive mental health (positive thoughts and feelings).

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Beauchet, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Beauchet O, Bastien T, Ho AHY, Vilcocq C, Galery K, Launay CP. Long-term effects of the Montreal museum of fine arts participatory activities on frailty in older community dwellers: results of the A-Health study. Eur Geriatr Med. 2021 Apr;12(2):295-302. doi: 10.1007/s41999-020-00408-w. Epub 2020 Oct 13. PMID 33051855
- [Derived] Beauchet O, Bastien T, Mittelman M, Hayashi Y, Hau Yan Ho A. Participatory art-based activity, community-dwelling older adults and changes in health condition: Results from a pre-post intervention, single-arm, prospective and longitudinal study. Maturitas. 2020 Apr;134:8-14. doi: 10.1016/j.maturitas.2020.01.006. Epub 2020 Jan 13. PMID 32143777